CLINICAL TRIAL: NCT05067673
Title: Association Between Tissue Changes in Lumbar Multifidae and Improvement in Pain and Disability After Dry Needling in Subjects With Nonspecific Low Back Pain. Randomized Clinical Trial.
Brief Title: Tissue Changes in Lumbar Multifidus After Dry Needling in Subjects With Nonspecific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Sebastián Rodríguez PosadaSebastián Rodríguez Posada, Principal investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 210108
Record Dates: First submitted 2021-09-14; First posted 2021-10-05 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain
Keywords: lower back pain; dry needling; ultrasound; disability
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind randomized clinical trial in parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo dry needling
  Interventions: Other: Placebo dry needling
- Experimental group (Experimental): Dry needling
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — The dry needling will be performed using disposable stainless steel needles (AGU-PUNT needles of size 0.30x50mm or 0.30x60mm depending on the patient) that will be inserted perpendicularly at the point of major hyperalgesia using the Hong technique. The patient will be in the prone position with a pillow placed in the abdominal region. The area will be cleaned with an antiseptic and allowed to air dry for 3 minutes. After this time, the needle will be inserted at the point indicated by the evaluator before reaching the lumbar multifidus by means of echolocation. Once it is assured that it is in the right place, a total of 10 repetitions are performed. The needle will be removed by depositing it in a needle container and a compression will be removed in the treated area until hemostasis is achieved.
  Arms: Experimental group
Other: Placebo dry needling — Placebo dry needling will be performed with DongBang DB100 Acupuncture Needles which, upon contact with the patient, retract, hiding in the needle handle. The patient will be in the prone position with a pillow in the abdominal region. The area will be cleaned with an antiseptic and allowed to air dry for 3 minutes. At the point indicated by the evaluator, the placebo needle will be placed initially and the introduction of the needle and its location will be simulated with the ultrasound system. 10 repetitions will be performed. The needle will be removed by depositing it in a needle container and a compression will be made in the treated area.
  Arms: Control group

SUMMARY:
Finding out if tissue changes (thickness, histogram and shrinkage rate) that occur in the lumbar multifidus after deep dry needling are related to changes in patient's pain and disability.

DETAILED DESCRIPTION:
Lower back pain in regarded as the main cause of disability in the world, which has a significant socio-economic impact. Deep dry needling is effective in handling such pain and is one of the techniques of choice by physiotherapists. In this area, the use of ultrasound provides information of interest such as length, thickness, diameter, cross-sectional area or muscle volume, among others.

Objective: Finding out if tissue changes (thickness, histogram and shrinkage rate) that occur in the lumbar multifidus after deep dry needling are related to changes in patient's pain and disability.

It's a double-blind randomized clinical trial in parallel groups. Patients will be randomly divided into 2 groups. One of them will receive dry needling and the other dry needling placebo. The initial, post-needling and a week after evaluations will be performed by a blinded to the intervention therapist.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Nonspecific pain in the lumbar region.

Exclusion Criteria:

* Previous surgery in the lumbosacral spine.
* Osteoporosis.
* Needle phobia.
* Neurogenic pain with positive tests or negative symptoms.
* Red flags: cauda equina syndrome, sudden weight loss, fracture, cancer, infection or systemic diseases.
* Pregnancy.
* Physiotherapy intervention in the 4 weeks prior to the intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in pain on the 10-point Visual Analog Scale (VAS, 0-10 score) at immediatelypost-needling and a week after. | Baseline, immediately post-needling and a week after.
  This scale shows concurrent and predictive validity in the assessment of pain. A difference of 2 points represents a clinically significant change that exceeds the limits of measurement error.

SECONDARY OUTCOMES:
Thickness of lumbar multifidus measured with Rehabilitive Ultrasound Imaging in millimeters | Baseline, immediately post-needling and a week after.
Histograms using image analysis | Baseline, immediately post-needling and a week after.
Pressure Pain threshold | Baseline, immediately post-needling and a week after.
  It will be measured by using a pressure algometer. Lumbar multifidus algometry is performed approximately 1.5 cm from the spinous process of the level to be evaluated. The measurement will be taken 3 times to avoid variability by instructing patients to say verbally when they begin to feel pain.
Disability | Baseline, immediately post-needling and a week after.
  it will be measured using the Roland-Morris questionnaire. Values range from 0 (absence of disability) to 24 (maximum level of disability).
Contraction time measured in milliseconds with M-mode | Baseline, immediately post-needling and a week after.
  The patient performs a hip extension in the prone position

CONTACTS AND LOCATIONS:
Locations (1):
- Sebastian, Torrejón de Ardoz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No